CLINICAL TRIAL: NCT00002290
Title: A Multi-Center, Double-Blind Trial to Evaluate the Safety and Efficacy of Concurrent Retrovir (Zidovudine) and Zovirax (Acyclovir) Therapy in Patients With Early Symptomatic Human Immunodeficiency Virus (HIV) Infection
Brief Title: The Safety and Effectiveness of Zidovudine Plus Acyclovir in Patients With Early HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 018A; 03
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-02

CONDITIONS: HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Drug Therapy, Combination; Acyclovir; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Opportunistic Infections; AIDS-Related Complex | interventions — Zidovudine; Acyclovir

INTERVENTIONS:
Drug: Zidovudine
Drug: Acyclovir

SUMMARY:
This double-blind, placebo-controlled study is designed to determine the long-term safety and efficacy of concurrent oral Retrovir / Zovirax (AZT and ACV) therapy and oral AZT therapy alone, in the treatment of early symptomatic HIV infection. Efficacy will be evaluated by monitoring the incidence, severity, and time of development of opportunistic infections and other manifestations of advanced symptomatic HIV infection. The effects of the combination and single AZT therapy on immune function and viral replication will also be evaluated. Study participants will be monitored for evidence of toxicity or intolerance to concurrent AZT / ACV administration and AZT therapy alone.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Early AIDS related complex (ARC).
* Willingness to be followed by the original study center for the duration of the trial (96 weeks).
* Ability to give informed consent.
* Patients may have associated lymphadenopathy (lymph nodes greater than or equal to 1 cm in two noncontiguous areas).

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Concurrent neoplasms other than basal cell carcinoma of the skin or in situ carcinoma of the cervix.
* Fever > 102 degrees F persisting for more than 14 consecutive days or more than 15 days in a 30-day interval, present at entry.
* Severe malabsorption (evidenced by persistent diarrhea of greater than 4 weeks duration with = or > 6 loose stools per day accompanied by significant weight loss).

Concurrent Medication:

Excluded:

* Acyclovir (ACV) therapy for chronic or recurrent herpes simplex.

Patients with an AIDS-defining indicator disease as outlined by the CDC surveillance definition for AIDS which includes opportunistic infections or neoplasms, HIV neurologic disease, AIDS dementia or the "wasting syndrome" are excluded.

Prior Medication:

Excluded within 4 weeks of study entry:

* Any other experimental therapy.
* Drugs which cause significant bone marrow suppression.
* Rifampin or rifampin derivatives.
* Cytolytic chemotherapy.
* Drugs which cause significant nephrotoxicity or hepatotoxicity.
* Immunomodulating agents, including steroids, interferon, Isoprinosine, immunoglobulin or interleukin 2.
* Excluded within 8 weeks of study entry:
* Antiretroviral agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Birmingham Veterans Administration Med Ctr / Univ of Alabama, Birmingham, Alabama
  - Univ of Arizona / Health Science Ctr, Tucson, Arizona
  - ViRx Inc, San Francisco, California
  - Georgetown Univ Med Ctr / Main Hosp 4, Washington D.C., District of Columbia
  - Veterans Administration Med Ctr, Bay Pines, Florida
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Harper Hosp, Detroit, Michigan
  - Univ of Pennsylvania / HIV Clinic, Philadelphia, Pennsylvania
  - Vanderbilt School of Medicine, Nashville, Tennessee
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Univ of Utah School of Medicine, Salt Lake City, Utah
  - Univ of Virginia Health Sciences Ctr, Charlottesville, Virginia
  - Richmond AIDS Consortium, Richmond, Virginia